CLINICAL TRIAL: NCT01217138
Title: Make up for the Epinephrine Autoinjector: Effect on Its Use by Untrained Users
Brief Title: Make up for the Epinephrine Autoinjector
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Gazi University Faculty of Medicine
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 232-05/25/2009
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2010-10-08 (Estimated); Status verified 2010-10

CONDITIONS: Anaphylaxis
Keywords: Anaphylaxis, autoinjector, design, epinephrine
MeSH Terms: conditions — Anaphylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Original epinephrine autoinjector group (Other): Participants were given original epinephrine autoinjector trainer wrapped by a gray sticky paper.
  Interventions: Device: Epinephrine autoinjector
- Modified epinephrine autoinjector group (Active Comparator): Participants were given the same epinephrine autoinjector trainer wrapped by a gray sticky paper which was modified by changing gray safety cap to red with an atomizer paint and placing a yellow arrow pointing to the black injection tip.
  Interventions: Device: Epinephrine autoinjector

INTERVENTIONS:
Device: Epinephrine autoinjector — We used 2 epinephrine autoinjector trainers and wrapped them by a gray sticky paper. Then,modified one of the trainers by changing gray safety cap to red with an atomizer paint and placing a yellow arrow pointing to the black injection tip.We provided three-step written and visual instruction sheet to use epinephrine autoinjector in Turkish same as given on the original trainer and changed that of the second trainer according to the modifications we made. Scoring system originally devised by Sicherer et al was used. Participants successively doing all steps were accepted to demonstrate autoinjector use correctly. Participants who tackled with black tip of autoinjector in order to eject needle after removing safety cap was regarded as unsuccessful since this may cause unintentional injection of epinephrine. All participants were scored and timed separately.
  Other Names: Epipen trainer®, Meridian Medical Technologies, Inc. Columbia, USA

SUMMARY:
Part of the problems related with proper use of epinephrine autoinjector may be related with the design of the autoinjector itself.The aim of the study is to investigate whether minor modifications in the design of currently available epinephrine autoinjector ease its use and abrogate common use errors.

DETAILED DESCRIPTION:
All interns except the ones who previously worked in allergy department in a medical school were invited to the study. Two identical epinephrine autoinjector trainers (Epipen trainer®) were used, one of which was modified by changing gray safety cap to red and placing a yellow arrow pointing to the black injection tip. Written and visual instruction sheet for each trainer was provided. Participants were asked to demonstrate the use of Epipen trainer either with the original or the modified one. They were scored and timed for demonstration. Primary study parameter was the rate of participants correctly demonstrating the use of epinephrine autoinjector. Secondary study parameters were the mean total score, mean time required to administer autoinjector and unintentional self injection of autoinjector into thumb.

ELIGIBILITY:
Inclusion Criteria:We invited all interns in our faculty to inform about the study and included the ones who gave informed consent -

Exclusion Criteria:Interns who previously worked in allergy department were excluded.

-

Ages: 21 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Rate of participants correctly demonstrating the use of epinephrine autoinjector.

SECONDARY OUTCOMES:
Mean total score participants get during demonstration of epinephrine autoinjector use
Mean time required to administer epinephrine autoinjector
Unintentional self injection of autoinjector into thumb

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Bakirtas, Principal Investigator — Gazi Universitry Faculty of Medicine, Department of Pediatric Allergy and Asthma; Mustafa Arga, Principal Investigator — Gazi Universitry Faculty of Medicine, Department of Pediatric Allergy and Asthma; Ferhat Catal, Principal Investigator — Gazi Universitry Faculty of Medicine, Department of Pediatric Allergy and Asthma; Oksan Derinoz, Principal Investigator — Gazi Universitry Faculty of Medicine, Department of Pediatric Emergency; Sadik M Demirsoy, Study Director — Gazi Universitry Faculty of Medicine, Department of Pediatric Allergy and Asthma; Ipek Turktas, Study Director — Gazi Universitry Faculty of Medicine, Department of Pediatric Allergy and Asthma

REFERENCES:
- [Derived] Bakirtas A, Arga M, Catal F, Derinoz O, Demirsoy MS, Turktas I. Make-up of the epinephrine autoinjector: the effect on its use by untrained users. Pediatr Allergy Immunol. 2011 Nov;22(7):729-33. doi: 10.1111/j.1399-3038.2011.01195.x. Epub 2011 Jul 13. PMID 21749463